CLINICAL TRIAL: NCT03679026
Title: The "Motoric Cognitive Risk" Syndrome in the Canadian Population: Analysis of Baseline Assessment of the Canadian Longitudinal Study on Aging (CLSA)
Brief Title: The "Motoric Cognitive Risk" Syndrome in the Canadian Population
Acronym: MCR-CardioV
Status: Active, not recruiting | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, Professor of Geriatrics, Jewish General Hospital
Other Study IDs: CODIM-FLP-16 261
Record Dates: First submitted 2018-08-21; First posted 2018-09-20 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Cognition Disorders in Old Age; Cardiovascular Diseases; Dementia
MeSH Terms: conditions — Cardiovascular Diseases; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CVRF: individuals with cardio-vascular risk factors and diseases
  Interventions: Other: Summarize of participants' characteristics using means and standard deviations or frequencies and percentages
- WCVRF: individuals without cardio-vascular risk factors and diseases
  Interventions: Other: Summarize of participants' characteristics using means and standard deviations or frequencies and percentages

INTERVENTIONS:
Other: Summarize of participants' characteristics using means and standard deviations or frequencies and percentages — Participants' baseline characteristics will be summarized using means and standard deviations or frequencies and percentages, as appropriate.

SUMMARY:
Cognition and locomotion are two human abilities controlled by the brain. Their decline is highly prevalent with aging, and is greater than the simple sum of their respective prevalence, suggesting a complex age-related interplay between cognition and locomotion. Recently, a systematic review and meta-analysis has provided evidence that poor gait performance predicts dementia and, in particular, has demonstrated that "motoric cognitive risk" (MCR) syndrome, which has been described in cognitively healthy individuals and combines subjective cognitive complaint with objective slow gait speed, is a pre-dementia syndrome. The uniqueness of "motoric cognitive risk" (MCR)syndrome is that it does not rely on a complex evaluation or laboratory investigations. Thus, it is easy to apply in population-based settings. The overall objective of the proposal is to examine the epidemiology of the newly reported "motoric cognitive risk" (MCR) syndrome, in the Quebec population using the database of the NuAge study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals eligible for this study will be participants of the NuAge study

Exclusion Criteria:

* Individuals not eligible for the NuAge study
* dementia
* mobility disability
* no information about cognitive complaint
* no measure of walking speed

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals eligible for this study will be participants of the comprehensive Canadian Longitudinal Study on Aging (n=30,097). They are separated in four age groups (i.e.; 45-54, 54-64, 65-74 and 75-85). Each group will be divided in two subgroups: individuals with and without cardio-vascular risk factors and diseases.
Sampling Method: Non-Probability Sample
Enrollment: 1461 (Estimated)
Dates: Start 2017-08-22 (Actual); Primary Completion 2021-08-21 (Actual); Study Completion 2024-12-21 (Estimated)

PRIMARY OUTCOMES:
Cardio-vascular risk factors and diseases assessed using reported health condition | 1 day
  medical history

SECONDARY OUTCOMES:
Cardio-vascular risk factors and diseases assessed using physical examination: BMI | 1 day
  body mass index
Cardio-vascular risk factors and diseases assessed using physical examination: HW ratio | 1 day
  hip-waist ratio
Cardio-vascular risk factors and diseases assessed using physical examination: blood pressure | 1 day
  (value of systolic, diastolic when participants are seated in an upright position in a chair)
Disability and functional limitations | 1 day
  Disability and functional limitations : ADL (activities of daily life)
Disability and functional limitations | 1 day
  Disability and functional limitations : IADL (instrumental activities of daily life)
Disability and functional limitations | 12 months
  History of falls during the past 12 months
Depression | 1 day
  measured by the 10 items of the Center for Epidemiological Studies Short Depression Scale. Participants with a score of 10 or greater are considered as depressed. Scores with more than 2 missing items will be excluded.
Cognitive performance | 1 day
  Prospective Memory Test (PMT)
Cognitive performance | 1 day
  Stroop Neurological Screening Test
Cognitive performance | 1 day
  Controlled Oral Word Association Test (FAS)
Cognitive performance | 1 day
  Choice Reaction Time Test (CRT)
physical and mental health | 1 day
  Number of drugs daily taken
physical and mental health | 1 day
  Self-perception of health and mental health
Physical performance | 1 day
  Muscle strength estimated using the handgrip strength
Physical performance | 1 day
  five-time sit-to-stand test
Physical performance | 1 day
  Physical Activity Scale for the Elderly, scored between 0 and 400, low scores indicate sarcopenia

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada